CLINICAL TRIAL: NCT04190173
Title: Efficacy of Prucalopride in Critically Ill Patients With Paralytic Ileus; a Pilot Randomized Double-blind Controlled Trial
Brief Title: Efficacy of PRUcalopride in Critically Ill Patients With Paralytic ILeus
Acronym: EPRUCIL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Panu Wetwittayakhlang, Principal investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 59-394-14-1
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Paralytic Ileus; Critically Ill
Keywords: Prokinetic; Prucalopride
MeSH Terms: conditions — Intestinal Pseudo-Obstruction; Critical Illness | interventions — prucalopride

STUDY DESIGN:
Intervention Model Description: Consecutive enrolment parallel group in intervention group and placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention was blinded to patients, nurse, investigators, and radiologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prucalopride (Experimental): Prucalopride (Trade name: Resolor) 2 mg oral or tube feeding once daily 5 consecutive days Decrease dose to 1 mg once daily in patient with end stage kidney disease or Cirrhosis Child Pugh C
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Placebo tablet to mimic Prucalopride made by starch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — 1-2 mg once daily enteral feeding for 5 consecutive days
  Other Names: Resolor
  Arms: Prucalopride
Drug: Placebo — 1/2-1 tablet once daily enteral feeding for 5 consecutive days
  Arms: Placebo

SUMMARY:
Paralytic ileus is a common intestinal dysfunction in critically ill patients. There are still no established the effective medications except correcting the primary causes and prokinetics trial which limited in efficacy and potential adverse events.

DETAILED DESCRIPTION:
Prucalopride, a highly selective 5-HT4 receptor agonist, accelerates gastrointestinal transit which may reduce severity of ileus. Furthermore, there is no report of serious cardiac and neurological side effects. We aim to evaluate the efficacy of prucalopride as a prokinetic of choice on paralytic ileus in critically ill patients.

ELIGIBILITY:
Inclusion:

* Medical patients with APACHE II score >= 15
* Paralytic ileus: small bowel diameter >= 4 cm or large bowel diameter >= 6 cm

Exclusion:

* no current prokinetic use
* Severe peritonitis or bowel inflammation
* ESRD needed hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Change of maximum bowel diameter from baseline at 24 hours | after first dose intervention to next 24 hours
  measure on plain abdominal radiography by blinded radiologist
Change of maximum bowel diameter from baseline at 48 hours | after first dose intervention to next 48 hours
  measure on plain abdominal radiography by blinded radiologist
Change of maximum bowel diameter from baseline at 72 hours | after first dose intervention to next 72 hours
  measure on plain abdominal radiography by blinded radiologist
Change of maximum bowel diameter from baseline at 96 hours | after first dose intervention to next 96 hours
  measure on plain abdominal radiography by blinded radiologist
Change of maximum bowel diameter from baseline at 120 hours | after first dose intervention to next 120 hours
  measure on plain abdominal radiography by blinded radiologist

SECONDARY OUTCOMES:
change of abdominal circumference from baseline at 24 hours | after first dose intervention to next 24 hours
  measured at umbilical level
change of abdominal circumference from baseline at 48 hours | after first dose intervention to next 48 hours
  measured at umbilical level
change of abdominal circumference from baseline at 72 hours | after first dose intervention to next 72 hours
  measured at umbilical level
change of abdominal circumference from baseline at 96 hours | after first dose intervention to next 96 hours
  measured at umbilical level
change of abdominal circumference from baseline at 120 hours | after first dose intervention to next 120 hours
  measured at umbilical level

CONTACTS AND LOCATIONS:
Overall Officials: Sawangpong Jandee, Dr., Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No